CLINICAL TRIAL: NCT01373333
Title: Use Of 3,4-Diaminopyridine (3,4-DAP) In The Treatment Of Lambert Eaton Myasthenic Syndrome
Acronym: 34-DAP
Status: No longer available | Type: Expanded Access
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 102,384; NCT00817856 (obsolete NCT alias)
Record Dates: First submitted 2011-06-13; First posted 2011-06-14 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Lambert-Eaton Myasthenic Syndrome
MeSH Terms: conditions — Lambert-Eaton Myasthenic Syndrome

INTERVENTIONS:
Drug: 3,4 DAP — Recommended maximum dosage: 20mg four times daily and if needed an additional 20 mg per day for a total of 100 mg per day. Drug must be kept refrigerated at all times.

SUMMARY:
Compassionate use of orphan drug 3,4-Diaminopyridine(DAP) in Treatment of Lambert Eaton Myasthenic Syndrome (LEMS). 3,4-DAP is used to decrease the muscle weakness associated with LEMS and hopefully will decrease the need for prednisone and all other therapies that were previously required to control symptoms. How long a patient will take 3,4 DAP depends upon if he/she is seeing benefits from the medication or experiencing side effects that will prevent them from continuation in the study.

DETAILED DESCRIPTION:
3,4-diaminopyridine (3,4-DAP) decreases symptoms of weakness in patients with LEMS, and therefore can be used to decrease the amount of immune modulation therapy needed to provide an equivalent degree of disease control.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of LEMS with or without any of the following: evidence of underlying malignancy, presence of P/Q or N-type calcium channel antibodies, electrodiagnostic evidence of a presynaptic defect of neuromuscular junction transmission.None of these laboratory findings are required for inclusion in this study.
2. P/Q and N type calcium channel antibodies are measured in the blood as a routine laboratory test during the course of initial diagnosis, but 10-20% of patients with LEMS do not have elevated levels of these antibodies.

Exclusion Criteria:

1. Hypersensitivity to any component of this medication.
2. History of past or current seizures.
3. History of asthma.
4. Evidence of prolonged QT syndrome. There is no absolute upper limit of normal for the QTc interval.
5. Family history of prolonged QTc syndrome, history of unexplained syncope, seizures or cardiac arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-09; Primary Completion 2012-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry H Levin, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States